CLINICAL TRIAL: NCT04974099
Title: Personalized Infliximab Induction Strategy With Model-informed Dosing in Patients With Crohn's Disease
Acronym: REMODEL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This was the Pilot study. The larger, confirmatory study has started
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-0282
Record Dates: First submitted 2021-06-29; First posted 2021-07-23 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: The intervention cohort includes patients, age 6-22 years old who have been diagnosed with CD, are naïve to anti-TNF medications and are scheduled to start infliximab (or infliximab biosimilar).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RoadMAB dashboard system (Experimental): The intervention includes utilizing Clinical and Patient Decision Support Software (RoadMABTM) that will guide the selection of the first infliximab dose followed by subsequent infliximab dose and dosing interval during the maintenance phase. During induction, three infusions will occur at 0, 2 and 6 weeks, respectively. The RoadMABTM dashboard will utilize PK modeling software to provide an infliximab starting dose recommendation (range of 5-12 mg/kg) based on the patients biochemical profile. As noted, dosing frequency (weeks) during induction will not be altered during this study. Following the first three doses, the clinician will be informed of their patients PK profile within the RoadMABTM program and with a shared document (paper). RoadMABTM will provide additional dosing recommendations after each infusion (based on the latest drug concentration measures and blood biomarkers) with the final dose and interval selected by the treating physician.
  Interventions: Device: RoadMAB; Drug: Precision dosing with a dashboard

INTERVENTIONS:
Device: RoadMAB — The RoadMAB Dashboard is a real-time decision support system that incorporates PK model-informed Bayesian estimation to provide precision dosing at the point of care.
  Other Names: Precision dosing with a dashboard
Drug: Precision dosing with a dashboard — The trial is testing whether precision dosing can more reliably achieve the targeted trough concentrations compared to standard dosing

SUMMARY:
Approximately 3 million people in the United States are living with inflammatory bowel disease, which includes Crohn's Disease, with many of those being young children and adolescents. Physicians need better ways to inform decisions on treatment.

The main reason for this research study is to determine if a computer program that formulates a dose based on a patient's blood testing results can better achieve the optimal drug level as compared to standard dosing.

DETAILED DESCRIPTION:
This is a Pilot study to evaluate safety, feasibility and efficacy of utilizing pharmacokinetic modeling to provide an individualized infliximab induction regimen in children and young adults with moderate to severe Crohn's disease. This clinical study is designed with the hypothesis that treatment regimens that account for individual (patient) drug clearance (pharmacokinetic modeling) will not only be safe and cost-effective, but also more effective in reducing intestinal inflammation than as-labeled dosing (ALD) regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form from the patient (≥18 years old) or from parent/legal guardian if patient is <18 years old.
2. Written informed assent form from patient ≥11 years old.
3. Age criteria: ≥6 years to ≤22 years of age.
4. Diagnosis of Crohn's Disease
5. Starting infliximab (or biosimilar)
6. Anti-TNF naïve (never received infliximab, adalimumab, golimumab, certolizumab or anti-TNF biosimilar)
7. Fecal calprotectin >250 µg/g or fecal lactoferrin >10 µg/g (up to 6 weeks prior to starting infliximab) or endoscopic evidence of active Crohn's disease (up to 90 days prior to starting infliximab)
8. wPCDAI >12.5 (up to 6 weeks) prior to the first infliximab infusion
9. Negative urine pregnancy test for ALL female subjects
10. Negative TB (tuberculosis) blood test

Exclusion Criteria:

1. Diagnosis of ulcerative colitis or inflammatory bowel disease-unspecified
2. Prior treatment with infliximab, adalimumab, certolizumab or golimumab (or anti-TNF biosimilar)
3. Active or prior evidence in past 12 months of internal (abdominal/pelvic) penetrating fistula(e)
4. Active intestinal stricture (luminal narrowing with pre-stenotic dilation >3mm), intra-abdominal abscess or perianal abscess
5. Active Clostridium difficile infection or other known bacterial/viral gastroenteritis in last two weeks
6. Current ileostomy, colostomy, ileoanal pouch, and/or previous extensive small bowel resection leading to short bowel syndrome
7. History of autoimmune disease (including autoimmune hepatitis, primary sclerosing cholangitis, thyroiditis, psoriasis or juvenile idiopathic arthritis)
8. Treatment with another investigational drug within four weeks.
9. Treatment with intravenous antibiotics within four weeks.
10. Planned continuation of 6-mercaptopurine or azathioprine (Imuran) during study.
11. Planned continuation of methotrexate during study.
12. Treatment with intravenous corticosteroids within two weeks.
13. Currently pregnant, breast feeding or plans in next 12 months to become pregnant
14. Inability or failure to provide informed assent/consent

Ages: 6 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Obtain safety data for optimal dosing strategy and sample size estimation | 2 years
  Number of adverse and/or serious adverse events
Enrollment feasibility | 2 years
  Evaluate the rate of recruitment
Completion feasibility | 2 years
  Number of patients that complete the study
Rate of patient adherence to stool and blood sample collections | 2 years
  patient adherence to stool and blood sample collections
RoadMAB Usability | 2 years
  Evaluate rate of physician adherence to RoadMAB dosing recommendation
RoadMAB Efficacy | 2 years
  Rate of achieving infus3 (Visit 4) infliximab concentration between 16-24 μg/ml as a dichotomous outcome

SECONDARY OUTCOMES:
Evaluate accuracy of infliximab concentration targets - Median difference infus3 | 2 years
  Median difference of infus3 (Visit 4) levels between cases and controls
Evaluate accuracy of infliximab concentration targets - Incidence | 2 years
  Incidence of achieving infus2 (Visit 3) level between target range of 26-34 μg/ml as a dichotomous outcome
Evaluate accuracy of infliximab concentration targets - Median difference infus2 | 2 years
  Median difference of infus2 (Visit 3) levels between cases and controls
Evaluate accuracy of infliximab concentration targets - Maintenance | 2 years
  Rates of achieving maintenance targets infus4-6 (Visits 5-7) between 5-10 μg/ml
Evaluate accuracy of infliximab concentration targets | 2 years
  Rate of development of antiinfliximab antibodies at any infusion between cases and controls
Infus4 (Visit 5) and infus6 (Visit 7): Clinical Response | 2 years
  Improvement in baseline wPCDAI by >17.5 or a wPCDAI<12.5
Infus4 (Visit 5) and infus6 (Visit 7): Clinical Remission | 2 years
  wPCDAI <12.5 and off corticosteroids
Sustained Remission | 2 years
  wPCDAI <12.5 and off prednisone for all visits from infus4 (Visit 5) to infus6 (Visit 7)
Infus4 (Visit 5) and Infus6 (Visit 7): Fecal Biochemical Response | 2 years
  ≥50% improvement in fecal calprotectin
Infus4 (Visit 5) and Infus6 (Visit 7): Fecal Biochemical Remission | 2 years
  fecal calprotectin <250 μg/g
Infus6 (Visit 7): Rate of transmural ileal | 2 years
  ileum subscore stage 0 (score = 0)
Infus6 (Visit 7): Rate of colonic healing | 2 years
  all segments of colon subscore stage 0 (score = 0)
Infus6 (Visit 7): Rate of total bowel healing | 2 years
  total ileum and colonic subscore is not greater than stage 0 on either individual score

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Minar, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No